CLINICAL TRIAL: NCT05436821
Title: INVESTIGATION OF THE EFFECT OF NONINVASIVE AURICULAR VAGUS NERVE STIMULATION ON PERFORMANCE IN PROFESSIONAL ATHLETES
Brief Title: The Effect of Vagus Nerve Stimulation on Sportive Performance.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: İSMAİL CEYLAN (Other)
Responsible Party: Sponsor-Investigator, İSMAİL CEYLAN, Head of hand therapy clinic. PhD., Ahi Evran University Education and Research Hospital
Organization: Ahi Evran University Education and Research Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12068451746
Record Dates: First submitted 2022-06-24; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Sports Performance
Keywords: Vagus, autonomic nerve system

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vagus nerve stimulation (Experimental): Auricular Vagus Nerve Stimulation (AVNS) was applied to the experimental group. AVNS application was applied to both ears simultaneously for 20 minutes, with waveform biphasic asymmetric, pulse duration 300 microseconds and frequency 25 hertz. AVNS application was made with Vagustim brand device.
  The acute effect of the application was evaluated in both groups by isometric quadriceps strength measurement, heart rate variability measurement, grip strength measurement and modified star balance test measurement performed before and after the single session AVNS.
  Interventions: Device: Auricular vagus nerve stimulation
- Control group (Sham Comparator): Sham Auricular Vagus Nerve Stimulation (AVNS) was applied to the experimental group. AVNS application was applied to both ears simultaneously for 20 minutes, with no pulse. AVNS application was made with Vagustim brand device.
  Before and after sham AVNS isometric quadriceps strength measurement, heart rate variability measurement, grip strength measurement and modified star balance test measurement performed.
  Interventions: Device: Sham Auricular Vagus Nerve Stimulation (AVNS)

INTERVENTIONS:
Device: Auricular vagus nerve stimulation — Autonomic nerve system regulation
  Arms: Vagus nerve stimulation
Device: Sham Auricular Vagus Nerve Stimulation (AVNS) — Sham Auricular Vagus Nerve Stimulation (AVNS)
  Arms: Control group

SUMMARY:
Performance is defined as the physiological potential required for an individual's physical activity. The sportive activity that he creates with his potential is defined as the sportive performance level of the individual. There are many factors that determine athletic performance. These factors are; environmental factors such as heredity, physical structure, training level, technical capacity and mental adequacy, quality of training areas, nutritional quality, suitability in weather conditions. All these factors affect the planning of multidisciplinary and interdisciplinary approaches that affect the performance of the athlete.

Autonomic regulation is very important for the reorganization of the athlete's performance. Auricular vagus nerve stimulation (VNS) is a non-invasive method. With this method, autonomic nervous system regulation can be done practically. In the literature, there are no studies examining the effect of VNS on recovery and performance in athletes.

DETAILED DESCRIPTION:
In this study, the effects of auricular vagus nerve stimulation on performance and recovery were investigated, which was designed as a randomized controlled trial, a single session of VSU was applied to 60 male professional athletes (30 experimantal, 30 control). The normal application waveform was biphasic asymmetric, with a pulse duration of 300 microseconds and a frequency of 25 hertz, for 20 minutes and continuously.

ELIGIBILITY:
Inclusion Criteria:

* Being an athlete who continues an active sports life.
* Not have an ongoing injury that prevents participation in the study
* To make a medium and high level weekly training period.

Exclusion Criteria:

* Having a systemic or neurological disease affecting the autonomic nervous system.
* Be younger than 18 years old and over 40 years old.
* Loss of sensation affecting the inner and outer ear, etc. have the disease.
* Having any acute systemic disease to exercise.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 60 people between the ages of 18-40, who applied to the Orthopedics and Traumatology Department of Private Ataşehir Florence Nightingale Hospital, performed pre-mid-end performance training, completed rehabilitation after injury, continued active sports life, and had moderate and high training tempo. male professional athlete.
Enrollment: 60 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Heart rate | 1 day
  Heart rate variability was controlled for autonomic measurement evaluation in both groups. Polar H7 heart rate sensor chest strap and wrist watch were used to measure analytical heart rate variability.

CONTACTS AND LOCATIONS:
Overall Officials: Adem Çalı, PhD, Principal Investigator — Bahçeşehir University
Locations (1):
- Kırşehir ahi Evran Üniversitesi, Kırşehir, Central Anatolia, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Calixtre LB, Oliveira AB, de Sena Rosa LR, Armijo-Olivo S, Visscher CM, Alburquerque-Sendin F. Effectiveness of mobilisation of the upper cervical region and craniocervical flexor training on orofacial pain, mandibular function and headache in women with TMD. A randomised, controlled trial. J Oral Rehabil. 2019 Feb;46(2):109-119. doi: 10.1111/joor.12733. Epub 2018 Oct 26. PMID 30307636
- [Derived] Caliota A, Ozden AV, Ceylan I. Effects of a single session of noninvasive auricular vagus nerve stimulation on sports performance in elite athletes: an open-label randomized controlled trial. Expert Rev Med Devices. 2024 Mar;21(3):231-237. doi: 10.1080/17434440.2023.2299300. Epub 2023 Dec 30. PMID 38146234